CLINICAL TRIAL: NCT00600418
Title: Identifying Posttraumatic Distress Among Toddlers and Their Parents Following Ongoing Exposure to Terrorism or War
Brief Title: Identifying Toddlers and Their Parents Who Are Suffering From Posttraumatic Distress Following War and Terror
Status: Completed | Type: Observational
Sponsor: Herzog Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ruth Pat-Horenzcyk, Director Children and Adolescents Clinical Services, Herzog Hospital
Other Study IDs: Rpat2CTIL
Record Dates: First submitted 2007-08-13; First posted 2008-01-25 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; DYADIC TREATMENT; WAR AND TERROR; Posttraumatic symptoms among toddlers
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The project is aimed at identifying children who are suffering from posttraumatic distress and increasing capacity to provide treatment for them and for their caretakers. The project will be implemented in 3 cities in Israel, Haifa, Kiryat Shmona and Sderot, exposed to terrorism and the effects of war

DETAILED DESCRIPTION:
A. Screening of young children and implementation of treatment The screening will consist of self-report questionnaires and a clinical interview with parents, conducted by trained professional about exposure to traumatic events and resulting post-traumatic specific symptoms among the toddlers and their parents. The screening procedure is bases on the accumulated clinical experience and empirical data gained in the ongoing similar project in Sderot. The level of cooperation by parents and teachers in the ongoing project has been exceptionally high, indicating a tremendous need for knowledge, skills and support. Based upon our previous experience, it is anticipated well-baby clinic nurses will also be extremely interested participation.

B. Workshops for parents, teachers, nurses The knowledge and skills of preschool teachers and nurses working in all our projects sights (well baby clinics, day care centers and kindergartens) as well as parents will be increased by providing training regarding the impact of war related trauma on preschool children. Workshops will better equip teachers, nurses and parents with knowledge about the emotional impact of trauma on young children and will increase the skills to help preschool children contain emotional distress as well as to help them in coping with the emotional consequences of trauma exposure.

C. Treatment Interventions All toddlers identified with posttraumatic distress will receive dyadic treatment focused on dealing with posttrauma. Dyadic treatment involving parents and children is aimed at increasing the attunement of parents to their toddlers and their needs in times of crises. Local practitioners in Sderot implementing this cutting-edge treatment received specialized training adjusted to the context of terror and trauma by a child trauma specialist from Mount Sinai Medical Center in New York.

D. Evaluation of treatment Evaluation of treatment efficacy (dyadic treatment) will be assessed by pre and post interviews that will be conducted by trained professionals with all parents participating in the dyadic treatments in each of the three cities

ELIGIBILITY:
Inclusion Criteria:

* Families with children between the age 1-6 years.
* Families living in Sderot, Kyriat Shmona and Haifa

Exclusion Criteria:

* Severe developmental problems

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Families with children between the age 1-6 years
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
PTSD and behavioral and emotional problems | April 2007- December 2008

SECONDARY OUTCOMES:
Maternal depression and PTSD | Aprol 2007- December 2008

OTHER OUTCOMES:
Maternal flexibility | April 2008- December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Pat-Horenczyk, Ph.d, Principal Investigator — Isreal Center for the Treatment of Psychotrauma; Ruth Pat-Horenczyk, Ph.D, Principal Investigator — The Israel Center for the Treatment of Psychotrauma
Locations (1):
- Isreal Center for the Treatment of Psychotrauma, Jerusalem, Israel